CLINICAL TRIAL: NCT02635295
Title: Mobile Cooperation During the Clinical Practicum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Camilla Strandell-Laine, Doctoral candidate, University of Turku
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 45/2014
Record Dates: First submitted 2015-12-02; First posted 2015-12-18 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Learning
Keywords: Clinical practicum; Nursing student; Nurse teacher; Mobile technology; Cooperation; Nurse competence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mobile cooperation (Experimental): Nursing student - nurse teacher mobile cooperation during the clinical practicum.
  Interventions: Behavioral: Mobile cooperation during the clinical practicum
- Standard cooperation (No Intervention): Nursing student - nurse teacher standard cooperation during the clinical practicum.

INTERVENTIONS:
Behavioral: Mobile cooperation during the clinical practicum — The intervention include (1) use of mobile application in nursing student - nurse teacher (NT) cooperation during the 5 weeks clinical practicum and (2) training at the beginning of the clinical practicum in the functions of the mobile application by the researcher.
  Students in the intervention group use mobile application for documentation of the terms of hours, learning diaries, objectives as well as mid-point and end-evaluation during the clinical practicum. NT and students have direct access to documents in the mobile application and to wireless communication regardless of time and place. The actions in the mobile application are automatically saved and shared between student and the NT.
  Arms: Mobile cooperation

SUMMARY:
The aim of this study is:

1. to evaluate the effectiveness of the nursing student - nurse teacher mobile cooperation (MC) during the clinical practicum,
2. to measure the usability of the mobile application.

The detailed research questions and hypothesis of this study are as follows:

1. What is the impact of MC on the nurse competence level of nursing students evaluated by work role, teaching-coaching and therapeutic interventions?

   H1: Nursing students' using MC will have a stronger change in the self-assessed level of nurse competence than those using standard cooperation (SC).

   H2: Nursing students' using MC will have higher level of nurse competence assessed by mentors after clinical practicum than those using SC.
2. What is the impact of MC on the clinical self-efficacy level of nursing students?

   H3: Nursing students' using mobile cooperation will have a stronger change in the self-assessed level of self-efficacy in clinical performance than those using standard cooperation.
3. What is the impact of mobile cooperation on the satisfaction level of nursing students evaluated by supervisory relationship, pedagogical atmosphere on the ward and the role of nurse teacher?

   H4: Nursing students' using mobile cooperation will have higher level of satisfaction with the supervisory relationship, pedagogical atmosphere on the ward and the role of nurse teacher after clinical practicum than those using standard cooperation.
4. What is the perceived usability of the mobile application by the intervention group?

The ultimate goal is to establish a modern, innovative solution for the nursing student - nurse teacher cooperation to support and facilitate the clinical learning of nursing students during the clinical practicum.

DETAILED DESCRIPTION:
The study takes place in surgical and internal medicine wards and related specialties and subspecialties in five academic hospitals of one hospital district in Finland.The setting of the study have similar learning environments and mentors.

The sample size was determined with power analysis and the target sample size is 50 subjects per group i.e. 100 in total.

All eligible student participants are identified from the student group lists and the employment service database (Jobstep) of the polytechnic.

Students are recruited by means of direct invitation at the polytechnic. The recruitment is continued until number of eligible participants desired is achieved. The mentors from the wards, supervising the students during the study, are informed of the study and recruited by direct invitations by the researcher.

Students in the intervention group use MC during the 5 week clinical practicum, while participants in the control group use SC.

ELIGIBILITY:
Inclusion Criteria:

1. pre-registration nursing student in one polytechnic undertaking nursing, midwifery or public health nursing degree programme,
2. at least second-year students,
3. entering a five week internal medicine or surgical clinical practicum at the participating hospital district,
4. entering the clinical practicum in spring term 2015,
5. access to a smartphone or tablet PC running iOS or Android OS.

Exclusion Criteria:

1. pre-registration nursing students undertaking critical care nursing degree program,
2. is unable to enter the clinical practicum in spring term 2015,
3. has not access to an appropriate smartphone or tablet PC,
4. is unwilling to provide consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Changes in students' nurse competence level measured with the NCS | Baseline, week 5
  Changes in students' self-assessed level of the nurse competence measured with the Nurse Competence Scale (NCS) at baseline (before the intervention) and week 5 (after the intervention). In addition, mentors assesses the nurse competence of students at 5 week with the NCS.

SECONDARY OUTCOMES:
Changes in students' clinical self-efficacy measured with the SECP | Baseline, week 5
  Changes in students' self-assessments of their own self-efficacy measured with the Self-Efficacy in Clinical Performance Scale at baseline (before the intervention) and week 5 (after the intervention).
Students' satisfaction to the clinical learning environment measured with the CLES+T at ward level | At the baseline
  Students' satisfaction with the supervisory relationship, pedagogical atmosphere on the ward and the role of nurse teacher is measured with the Clinical Learning Environment, Supervision and Nurse Teacher Scale (CLES Scale) at ward level
Students' satisfaction to the clinical learning environment measured with the CLES+T2 at student level | Week 5
  Students' satisfaction with the supervisory relationship, pedagogical atmosphere on the ward and the role of nurse teacher is measured with the Clinical Learning Environment, Supervision and Nurse Teacher Scale (CLES+T2 Scale) at student level
Process evaluation by the students in the intervention group | Week 5, week 6, week 16
  The perceived usability of the mobile application is measured by the students with the System Usability Scale, SUS. The intervention is assessed by a structured process evaluation questionnaire at week 5 (after the intervention). The perceived effects and development propositions for the intervention are measured qualitatively at week 6 by a focus group interview (semi-structured questions) with students and at week 16 by student essays (open-ended questions).

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Strandell-Laine, PhD(c), Principal Investigator — University of Turku
Locations (1):
- University of Turku, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Strandell-Laine C, Saarikoski M, Loyttyniemi E, Meretoja R, Salminen L, Leino-Kilpi H. Effectiveness of mobile cooperation intervention on students' clinical learning outcomes: A randomized controlled trial. J Adv Nurs. 2018 Jun;74(6):1319-1331. doi: 10.1111/jan.13542. Epub 2018 Mar 6. PMID 29444335